CLINICAL TRIAL: NCT01321775
Title: Bevacizumab and Trastuzumab With Paclitaxel on Women With Her2+ Breast Cancer Weekly Paclitaxel Followed, After Surgery, by Encapsuled Liposomal Doxorubicin, Cyclophosphamide and Trastuzumab as Adjuvant Treatment After Surgery on Women With Her2+ Breast Cancer
Brief Title: Bevacizumab and Trastuzumab With Weekly Paclitaxel Followed, After Surgery, by Encapsuled Liposomal Doxorubicin, Cyclophosphamide and Trastuzumab as Adjuvant Treatment After Surgery on Women With Her2+ Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario Madrid Sanchinarro (Other)
Responsible Party: Sofia Perea, Fundación Hospital de Madrid
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVANTHER
Record Dates: First submitted 2011-03-23; First posted 2011-03-24 (Estimated); Last update posted 2011-03-24 (Estimated); Status verified 2010-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bevacizumab,Trastuzumab,Paclitaxel,Cyclophosphamide,Myocet (Experimental)
  Interventions: Drug: Bevacizumab,Trastuzumab,Paclitaxel,Cyclophosphamide,Myocet

INTERVENTIONS:
Drug: Bevacizumab,Trastuzumab,Paclitaxel,Cyclophosphamide,Myocet — Neo-adjuvant doses (12 weeks):
  Bevacizumab: 15mg/Kg every 3 weeks Trastuzumab: 4 mg/Kg (First dose) - 2mg/Kg every week. Paclitaxel: 80mg/m2 every week.
  Adjuvant doses:
  Trastuzumab: 8mg/Kg(first dose)- 6mg/Kg every 3 weeks (At least 9 months) Cyclophosphamide: 600mg/m2 every 3 weeks (9 months) Doxorubicin Liposomal: 50mg/m2 every 3 weeks (3 months)

SUMMARY:
The purpose of this study is to determine the efficacy of the combined therapy Bevacizumab, trastuzumab and paclitaxel in neo-adjuvant therapy in patients with breast cancer HER 2+ followed by surgery and adjuvant therapy (Cyclophosphamide, Trastuzumab and Doxorubicin liposomal).

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years
* Pre or post menopause patient with histology confirmation of breast cancer status II or III, Her2+ confirmed by FISH technique.
* Lesion bigger than 2cm.
* life expectancy > 12 weeks.
* Normal Heart function (LVEF>55%)
* Patient should give his/her signed, written informed consent.

Exclusion Criteria:

* Previous chemotherapy treatment.
* Previous treatment with HER2 or VEGF inhibitors.
* Pulmonary disease not controlled.
* Hypertension not controlled (systolic > 150 mmHg and/or diastolic > 100 mmHg) or significant cardiovascular disease (CVA/cerebral hemorrhage (6 months before inclusion), myocardial infarction (6 months before inclusion), unstable angina, congestive cardiac disease ≥ NYHA 2, or serious cardiac arrhythmia requiring medication.
* Antecedents of coagulopathy or clinically significant thrombosis.
* Major surgery, open biopsy or significant trauma 28 days before the inclusion in the study or planned major surgery during the study.
* Peripheral Neuropathy > CTC 2 at inclusion.
* Altered renal function a. Creatinine > 2.0 mg/dL or 177 mmol/L. b.Proteinuria > 2+ with reactive stick(dipstick). If screening proteinuria 2+, collection of 24h urine must show a value of proteins of 1 g/24h.
* Daily chronic treatment with corticosteroids
* Daily chronic treatment with aspirin (> 325 mg/day) o clopidogrel (> 75 mg/day)
* Antecedents or heritage evidence of bleeder diathesis or coagulopathy with risk of hemorrhage.
* Antecedents of abdominal fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months previous to the inclusion.
* Active infection to be treated with iv antibiotics
* Serious injury not curing, peptic ulcer or bone fracture.
* Pregnant or active sexual patient not using contraceptive methods. or lactating woman
* Current or recent treatment with another IMP or participation in another clinical trial (30 days before inclusion)
* Another primary tumor (including primary brain tumors)within 5 years to the study inclusion, apart from in situ cervix carcinoma, skin squamous carcinoma, both if they are appropriately treated, or skin basal cell cancer if controlled.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2009-08; Primary Completion 2013-02 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Pathologic response in breast and axilla | 16 weeks average

SECONDARY OUTCOMES:
To evaluate tumor markers as potential predictors of the pathologic response | baseline and 16 weeks average

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Hospital Ramón Y Cajal, Madrid, Madrid
  - Hospital Universitario, Madrid, Madrid
  - Complejo Hospital Costa Del, Marbella, Malaga